CLINICAL TRIAL: NCT01376115
Title: Drug Use Investigation for ARRANON G (Nelarabine) Injection 250mg
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: 112279
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — nelarabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects administered nelarabine: Subjects with T-cell acute lymphocytic leukemia (T-ALL) or T-cell lymphoblastic lymphoma (T-LBL) prescribed nelarabine during study period
  Interventions: Drug: Nelarabine

INTERVENTIONS:
Drug: Nelarabine

SUMMARY:
To investigate safety and efficacy on Japanese subjects treated with nelarabine injection for intravenous use in clinical settings of the following diseases:

1. T-cell acute lymphocytic leukemia (T-ALL)
2. T-cell lymphoblastic lymphoma (T-LBL) Also, "any adverse events involving neurological disorder, hypotension, and blood disorder and their details" are to be investigated as an item of particular concern. In addition, subject outcome (alive or dead) at one year after the start of treatment will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T-cell acute lymphocytic leukemia (T-ALL) or T-cell lymphoblastic lymphoma (T-LBL)

Exclusion Criteria:

* Subjects with hypersensitivity to nelarabine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with the following diseases in Japanese adults and children
  1. T-cell acute lymphocytic leukemia (T-ALL)
  2. T-cell lymphoblastic lymphoma (T-LBL)
Sampling Method: Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2008-01-18 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
The number of adverse events in Japanese subjects treated with nelarabine based on prescribing information under the conditions of general clinical practice. | 1 year
Any incidence of adverse events related to neurological disorder, hypotension, and blood disorder and their details | 1 year

SECONDARY OUTCOMES:
Outcome (alive or dead) at one year after the start of treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- University of Tsukuba Hospital, Tsukuba, Japan